CLINICAL TRIAL: NCT04071730
Title: Effects of Immulina Dietary Supplementation on Innate and Adaptive Immune Measures in Normal Human Volunteers
Brief Title: Effects of Immulina on Immune Measures
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mississippi Medical Center (Other)
Responsible Party: Principal Investigator, Gailen D. Marshall Jr., MD PhD, The R. Faser Triplett, Sr., MD Chair of Allergy and Immunology, Professor of Medicine, Pediatrics, Pathology and Population Science, University of Mississippi Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: 2019-0183
Record Dates: First submitted 2019-08-26; First posted 2019-08-28 (Actual); Last update posted 2022-05-19 (Actual); Status verified 2022-05

CONDITIONS: Effects of Immulina on Natural Killer Cells
Keywords: Immulina; Natural Killer Cells (NK); Dietary supplementation
MeSH Terms: interventions — Immulina

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immulina Dietary Supplementation (Experimental): Immulina Dietary Supplementation - 200 mg capsules; 800 mg/day; 2 (200 mg) capsules given by mouth in the morning and 2 (200 mg) capsules given by mouth in the evening for 4 weeks duration
  Interventions: Dietary Supplement: Immulina Dietary Supplementation
- Placebo (Placebo Comparator): Placebo - inert capsules; 2 capsules given by mouth in the morning and 2 capsules given by mouth in the evening for 4 weeks duration
  Interventions: Dietary Supplement: Immulina Dietary Supplementation

INTERVENTIONS:
Dietary Supplement: Immulina Dietary Supplementation — Immulina Dietary Supplementation is a highly standardized extract derived from various preparations of Spirulina, a cyanobacterium, marketed as a dietary supplement and has been utilized in several clinical studies describing its immunopotentiating properties.
  Other Names: Immulina; Spirulina

SUMMARY:
This small, randomized, double blind, placebo controlled pilot study is aimed at determining the effects of oral Immulina dietary supplementation on specific immune biomarkers in the blood.

DETAILED DESCRIPTION:
This small, randomized, double blind, placebo controlled pilot study is aimed at determining the effects of four weeks of daily Immulina dietary supplementation (800 mg/day) versus four weeks of daily placebo on natural killer (NK) cell numbers and/or natural killer (NK) cell activity in human peripheral blood mononuclear cells collected from human research participants who meet the trial's inclusion/exclusion criteria.

ELIGIBILITY:
Inclusion Criteria:

* Normal, generally healthy adults between ages 18-64 and who may or may not have a controlled disease(s). Examples of controlled diseases are controlled Type-2 diabetes mellitus, controlled hypertension, controlled allergic rhinitis, etc.

Exclusion Criteria:

* Individuals with specific disease entities, which, in the opinion of the Principal Investigator, could reasonably be assumed to have dysfunctional immune function as a component of their illness. These include HIV, AIDS, uncontrolled asthma, uncontrolled eczema, uncontrolled allergic rhinitis, uncontrolled urticaria, rheumatoid arthritis, lupus, inflammatory bowel disease, multiple sclerosis, Type-1 diabetes mellitus, Guillain-Barre syndrome, psoriasis, Grave's disease, Hashimoto's thyroiditis, myasthenia gravis or vasculitis.
* Individuals taking specific dietary supplements including probiotic, microalgae or beta glucan containing dietary supplements, fermented food products (such as yogurt, bean curd, etc.). If the potential participants reports usage of any of these products, they will be asked if they would be willing to withhold products for 30 days and then be re-screened for inclusion/exclusion criteria.
* Individuals who are unwilling to refrain for the duration of the trial from taking the specific dietary supplements and fermented food products including probiotic, microalgae or beta glucan containing dietary supplements, fermented food products (such as yogurt, bean curd, etc.).
* Pregnant females (because baseline immune responses, are altered by pregnancy)
* Individuals unable to speak, understand and read English

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-03 (Actual); Primary Completion 2021-02-28 (Actual); Study Completion 2021-03-11 (Actual)

PRIMARY OUTCOMES:
Natural Killer (NK) cell count | 4 weeks
  Differences in NK cell counts from baseline to 4 weeks

SECONDARY OUTCOMES:
Natural Killer (NK) cell cytotoxic activity | 4 weeks
  Differences in NK cell cytotoxic activity from baseline to 4 weeks
Cytokine profiles | 4 weeks
  Differences in in-Vitro peripheral blood mononuclear cell (PBMC) culture supernatants' cytokine profiles from baseline to 4 weeks (IFN-α, IFN-γ, IL-1β, IL-2, IL-4, IL-6, Il-10, IL-12, Il-15 and TNFα)
Immune cell populations | 4 weeks
  Differences in immune cell populations in PBMC from baseline to 4 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Gailen D Marshall, Jr., MD, PhD, Principal Investigator — Study Principal Investigator
Locations (1):
- University of Mississippi Medical Center, Jackson, Mississippi, United States

IPD SHARING:
Plan to Share IPD: No